CLINICAL TRIAL: NCT03789344
Title: Randomized Controlled Trials of Electro-acupuncture Effects on Perioperative Anxiety in Patients Treated With PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huan Wang, MD (Other)
Responsible Party: Sponsor-Investigator, Huan Wang, MD, director, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 301FW
Record Dates: First submitted 2018-12-24; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Percutaneous Coronary Intervention
Keywords: acupuncture, PCI
MeSH Terms: interventions — Acupuncture Therapy; Psychotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture treatment (Experimental)
  Interventions: Other: acupuncture
- Psychotherapy (Active Comparator)
  Interventions: Other: Psychotherapy
- blank control (Placebo Comparator)
  Interventions: Other: blank control

INTERVENTIONS:
Other: acupuncture — Acupuncturists apply the seven-days' electro-acupuncture treatment on the acupoints of Neiguan points and Daling points for 30min per day.
  Arms: Acupuncture treatment
Other: Psychotherapy — Subjects in psychotherapy group would be accepted 20mins- psychotherapy per day.
  Arms: Psychotherapy
Other: blank control — Blank control subjects would be observed only during this investigation.
  Arms: blank control

SUMMARY:
Randomized Controlled Trials of Electro-acupuncture Effects on Perioperative Anxiety in Patients Treated with PCI

ELIGIBILITY:
Inclusion Criteria:

* The main inclusion criteria were patients who underwent coronary angiography. Patients suffer from Generalized anxiety disorder(GOD).

Exclusion Criteria:

* The exclusion criteria were as follows: patients with chronic renal failure, chronic liver disease, bone disorders, and/or thyroid disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Heart Rate Variability at 7 days | at 1day before and 7 days after percutaneous coronary intervention
  The primary efficacy variable was the heart rate variability of patients accepted the PCI treatment between control group

SECONDARY OUTCOMES:
Scores of HAM-A | 1day before, 7，14 days after the intervene
  scores of HAM-A were recorded on 1day before, 7，14 days after the intervene
Scores of AIS | 1day before, 7，14 days after the intervene
  scores of AIS were recorded on 1day before, 7，14 days
Scores of HRSD | 1day before, 7，14 days after the intervene
  scores of HRSD were recorded on 1day before, 7，14 days

OTHER OUTCOMES:
inflammation mediators level in blood | 1day before, 7days after the intervene
  the blood level of IL-6 and Hs-CRP were detected

CONTACTS AND LOCATIONS:
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Pei JH, Gan F, Bai YH, Xing YL, Jia JJ, Wang H. Instant and short-term effects of acupuncture for depression and anxiety in unstable angina pectoris patients with percutaneous coronary interventions. Front Cardiovasc Med. 2024 Jan 19;11:1173080. doi: 10.3389/fcvm.2024.1173080. eCollection 2024. PMID 38312234